CLINICAL TRIAL: NCT03853772
Title: The Johns Hopkins Heartburn Center Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00201157
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Gastroesophageal Reflux Disease; Barrett Esophagus; Laryngopharyngeal Reflux; Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus; Laryngopharyngeal Reflux; Esophagitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multi-center, multi-year registry of patients with gastroesophageal reflux disease (GERD) undergoing diagnostic evaluation and/or treatment of GERD and associated diseases and complications.

DETAILED DESCRIPTION:
This registry is a prospective, multicenter registry of patients undergoing diagnostic evaluation and/or treatment of gastroesophageal reflux disease and associated diseases and complications.

Patients who are eligible will have disease and therapy-specific data collected throughout treatment and long-term (5-year) follow-up.

Electronic data capture via REDCap will be utilized for all sites.

ELIGIBILITY:
Inclusion Criteria:

* Referred GERD patients willing to participate in long term follow-up (5 years)

Exclusion Criteria:

* Potential participants will be excluded if unwilling or unable to complete surveillance questionnaires through this registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred by physicians having diagnostic evaluation or treatment for GERD.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-04-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Demographic and clinical data obtained via chart review and questionnaires | 5 years
  Establish a registry with collected data related to patients undergoing diagnostic evaluation and treatment of GERD and its associated diseases in multiple academic and community settings.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Canto, MD, Principal Investigator — Johns Hopkins University
Locations (9):
- United States (9):
  - UCI-Irvine, Orange, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - UNRMed-University of Nevada, Reno, Reno, Nevada
  - Weill Cornell, New York, New York
  - Geisinger, Danville, Pennsylvania
  - The Matagorda Regional Medical Group, Bay City, Texas
  - UT Health, Houston, Texas
  - Fox Valley Surgical Associates, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Research projects will be submitted to host (currently JHU) and accepted project will be granted access to read only de-identified database.
Supporting Information: Study Protocol, ICF
Time Frame: minimum 6 years
Access Criteria: Project submission to PI and or Heartburn Registry management team then if project accepted, security clearance and enrollment in REDCap and tutorial completions.